CLINICAL TRIAL: NCT02381418
Title: Immunogenicity, Reactogenicity and Safety of the Trivalent Influenza Subunit Vaccine Influvac® for the Southern Hemisphere Season 2015. An Open-Label, Baseline-Controlled Study in Two Age Groups: Adult Subjects ≥ 18 and ≤ 60 Years and Elderly Subjects ≥ 61 Years of Age
Brief Title: Annual Study to Investigate Inactivated Subunit Influenza Vaccine Due to New Virus Strains for the Southern Hemisphere 2015 Season
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INFL3014
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Committee for Medicinal Products for Human Use (CHMP) criteria
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Trivalent influenza subunit vaccine Influvac. "3x 15mcg Hemagglutinin Antigen (HA) per 0.5 ml,trivalent one injection at Day 1 "
  Interventions: Biological: Trivalent influenza subunit vaccine Influvac

INTERVENTIONS:
Biological: Trivalent influenza subunit vaccine Influvac — "3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1 "

SUMMARY:
Influenza (flu) viruses change continuously, therefore also the parts of viruses used in influenza vaccines can vary from year to year. The current study is a phase III A clinical trial with a commercially available vaccine (Influvac®) supplied in pre filled syringes. The objective of this study is to investigate the immunogenicity and safety and tolerability of the changed influenza vaccine virus composition in two groups of subjects in good health: subjects aged >= 18 and <= 60 years and subjects >= 61 years of age (elderly).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent and able to adhere to all protocol required study procedures.
* Men and women aged ≥ 18 and ≤ 60 years or ≥ 61 years of age at the day of study vaccination.
* Being in good health as judged by medical history, physical examination (if needed) and clinical judgment of the Investigator

Exclusion Criteria:

* Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
* A serious adverse reaction after a previous (influenza) vaccination.
* Presence of any significant condition that may prohibit inclusion as determined by the investigator.
* Seasonal or pandemic influenza vaccination or laboratory confirmed seasonal or pandemic influenza infection within the previous six months before study vaccination or planned vaccination during the study period.
* A history of Guillain-Barré syndrome or active neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Facility ID ORG-001075, Maroubra, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Influvac: Trivalent influenza subunit vaccine Influvac. "3x 15mcg Hemagglutinin Antigen (HA) per 0.5 ml,trivalent one injection at Day 1 "
Period: Overall Study
Arm/Group | Influvac
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Influvac: Trivalent influenza subunit vaccine Influvac. "3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1 "
Arm/Group | Influvac
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 71
  >=65 years | 48
Age, Continuous [Mean (Full Range); unit: years]
  adult (18-60 year old) | 41.2 [18 to 60]
  elderly adult (>=61 year old) | 71.5 [61 to 88]
Gender [Count of Participants; unit: Participants]
  Female | 58
  Male | 62
Region of Enrollment [Number; unit: participants]
  Australia | 120

OUTCOME MEASURES:

1. Primary Outcome: the Serum Antihemagglutinin Antibody Titers and the Derived Parameters Defined in the Committee for Medicinal Products for Human Use (CHMP) Note for Guidance on Harmonization of Requirements for Influenza Vaccines for Influenza Vaccines.
Description: Seroprotection and Seroconversion Rate for A/H1N1, A/H3N2, and B Strains 3 weeks After Vaccination in non-elderly adults and elderly adults.
Time Frame: 3 weeks post vaccination
Population: Two subjects were excluded from the efficacy sample due to major protocol violations with a potential effect on immunogenicity outcome.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Influvac
Number analyzed (Participants) | 118
percentage of subjects
  Percentage adults with seroprotection for A/H3N2 | 96.6 [88.3 to 99.6]
  Percentage adults with seroprotection for A/H1N1 | 96.6 [88.3 to 99.6]
  Percentage adults with seroprotection for B | 93.2 [83.5 to 98.1]
  Percentage elderly with seroprotection for A/H3N2 | 98.3 [90.9 to 100]
  Percentage elderly with seroprotection for A/H1N1 | 88.1 [77.1 to 95.1]
  Percentage elderly with seroprotection for B | 64.4 [50.9 to 76.4]
  Percentage adults with seroconversion for A/H3N2 | 83.1 [71.0 to 91.6]
  Percentage adults with seroconversion for A/H1N1 | 50.8 [37.5 to 64.1]
  Percentage adults with seroconversion for B | 52.5 [39.1 to 65.7]
  Percentage elderly with seroconversion for A/H3N2 | 76.3 [63.4 to 86.4]
  Percentage elderly with seroconversion for A/H1N1 | 32.2 [20.6 to 45.6]
  Percentage elderly with seroconversion for B | 35.6 [23.6 to 49.1]

2. Primary Outcome: the Serum Antihemagglutinin Antibody Titers and the Derived Parameters Defined in the Committee for Medicinal Products for Human Use (CHMP) Note for Guidance on Harmonization of Requirements for Influenza Vaccines for Influenza Vaccines.
Description: Mean fold increase in HI antibody titer 3 weeks After Vaccination in non-elderly adults and elderly adults.
Time Frame: 3 weeks post vaccination
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: fold change
Groups:
- Influvac: Trivalent influenza subunit vaccine Influvac. "3x 15mcg Hemagglutinin Antigen (HA) per 0.5 ml,trivalent one injection at Day 1 "
  Trivalent influenza subunit vaccine Influvac: "3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1 "
Arm/Group | Influvac
Number analyzed (Participants) | 118
fold change
  Mean fold increase A/H3N2 titer in adults | 19.2 [12.4 to 29.7]
  Mean fold increase A/H1N1 titer in adults | 8.6 [5.0 to 15.0]
  Mean fold increase B titer in adults | 5.7 [3.9 to 8.3]
  Mean fold increase A/H3N2 titer in elderly | 12.2 [8.3 to 17.8]
  Mean fold increase A/H1N1 titer in elderly | 3.1 [2.3 to 4.2]
  Mean fold increase B titer in elderly | 2.7 [1.9 to 3.8]

3. Secondary Outcome: Safety (Unsolicited Adverse Events) and Tolerability (Reactogenicity and Overall Inconvenience) of Influvac®.
Time Frame: up to 3 weeks post vaccination
Measure: Number; unit: participants
Arm/Group | Influvac
Number analyzed (Participants) | 120
participants
  Redness (18-60 years of age) | 6
  Swelling (18-60 years of age) | 5
  Itching (18-60 years of age) | 4
  Warmth (18-60 years of age) | 5
  Tenderness (18-60 years of age) | 22
  Pain (18-60 years of age) | 7
  Impairment of movement of arm (18-60 years of age) | 4
  Induration (hardening) (18-60 year of age) | 4
  Ecchymosis (blue spots) (18-60 year of age) | 0
  Fever >=38c (18-60 year of age) | 0
  Increased sweating (18-60 year of age) | 4
  Headache (18-60 year of age) | 10
  Malaise (18-60 year of age) | 5
  Fatigue (18-60 year of age) | 10
  Shivering (18-60 year of age) | 2
  Redness (>=61 year of age) | 0
  Swelling (>=61 year of age) | 1
  Itching (>=61 year of age) | 0
  Warmth (>=61 year of age) | 5
  Tenderness (>=61 year of age) | 7
  Pain (>=61 year of age) | 0
  Impairment of movement arm (>=61 year of age) | 0
  Induration (hardening) (>=61 year of age) | 1
  Ecchymosis (blue spots) (>=61 year of age) | 1
  Fever >-38c (>=61 year of age) | 1
  Increased sweating (>=61 year of age) | 2
  Headache (>=61 year of age) | 8
  Malaise(>=61 year of age) | 6
  Fatigue (>=61 year of age) | 9
  Shivering | 2

ADVERSE EVENTS:
Arm/Group | Influvac
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 19/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influvac (N=120)
vaccine site pain (General disorders) | 7 (9)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
application site pruritus (General disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fatigue (General disorders) | 3 (3)
malaise (General disorders) | 3 (3)
vaccination site warmth (General disorders) | 3 (3)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 2 (2)
respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other